CLINICAL TRIAL: NCT06268834
Title: Is Long-Term Proton Pump Inhibitor Use a Cause of Leaky Gut Syndrome: A Cross-Sectional Case-Control Study
Brief Title: Is Long-Term Proton Pump Inhibitor Use a Cause of Leaky Gut Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semih Sezer, clinic physician, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZonulinPPI
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Proton Pump Inhibitor Adverse Reaction
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using PPI (Experimental): Group receiving a long-term PPI (omeprazole, lansoprazole, pantoprazole, esomeprazole and rabeprazole) every day for at least 6 months or at least twice a week for at least 2 years.
  Interventions: Diagnostic Test: Blood for zonulin level was drawn from the group.
- Control (Experimental): A control group was formed from individuals who had never used PPI.
  Interventions: Diagnostic Test: Blood for zonulin level was drawn from the group.

INTERVENTIONS:
Diagnostic Test: Blood for zonulin level was drawn from the group. — Serum zonulin levels were determined by taking 5 cc blood from the antebrachial veins of the patients.

SUMMARY:
Our study aims to investigate the effect of bacterial overgrowth induced by long-term PPI use on zonulin levels.

DETAILED DESCRIPTION:
The study included a total of 75 participants, with 45 individuals classified as long-term PPI users and 30 as non-PPI users. The PPI user group was defined as those who had been consistently using PPIs (specifically omeprazole, lansoprazole, pantoprazole, esomeprazole, or rabeprazole) on a daily basis for a minimum of 6 months or at least twice a week for a minimum of 2 years. The control group comprised individuals who had never used PPIs. Venous blood samples were taken from all participants to measure serum zonulin levels.

ELIGIBILITY:
Inclusion Criteria:

The patient group was patients taking long-term PPIs (omeprazole, lansoprazole, pantoprazole, esomeprazole and rabeprazole) every day for at least 6 months or at least twice a week for at least 2 years.

A control group was formed from individuals who had never used PPI.

Exclusion Criteria:

Those with inflammatory bowel disease, celiac disease, type 1 diabetes, active gastroenteritis, acute kidney failure, chronic kidney failure, and those who had used antibiotics for any reason in the last 3 months, as well as those receiving probiotic drug support, were not included in the study

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Zonulin levels in long-term proton pump inhibitor users | Blood was drawn and collected during the examination and studied collectively after 3 months
  Approximately 5 cc of blood was drawn from the antebrachial veins of the patients to determine serum zonulin levels. Serum örnekleri -80 santigrat derecede 3 ay süreyle saklanmıştır. Serum örneklerindeki Zonulin seviyeleri Shanghai Crystal Day Biotech Co, Ltd, Shanghai, Çin'den ticari BT-LAB Human Zonulin ELISA kitleri (Kat. No. E1117Hu) kullanılarak ölçülmüştür. The test range of the kit was 2-600 ng/ml. The sensitivity of the test was 1.09 ng/ml. A serum zonulin level above 12 ng/ml was considered positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fasano A, Shea-Donohue T. Mechanisms of disease: the role of intestinal barrier function in the pathogenesis of gastrointestinal autoimmune diseases. Nat Clin Pract Gastroenterol Hepatol. 2005 Sep;2(9):416-22. doi: 10.1038/ncpgasthep0259. PMID 16265432
- [Background] El Asmar R, Panigrahi P, Bamford P, Berti I, Not T, Coppa GV, Catassi C, Fasano A. Host-dependent zonulin secretion causes the impairment of the small intestine barrier function after bacterial exposure. Gastroenterology. 2002 Nov;123(5):1607-15. doi: 10.1053/gast.2002.36578. PMID 12404235
- [Background] Haastrup PF, Thompson W, Sondergaard J, Jarbol DE. Side Effects of Long-Term Proton Pump Inhibitor Use: A Review. Basic Clin Pharmacol Toxicol. 2018 Aug;123(2):114-121. doi: 10.1111/bcpt.13023. Epub 2018 May 24. PMID 29658189